CLINICAL TRIAL: NCT06268054
Title: A National, Multicenter, Randomized, Double-blind, Phase III, Crossover Clinical Trial to Assess the Efficacy and Safety of DEH113 in the Treatment of Menstrual Cramp Pain Associated With Primary Dysmenorrhea.
Brief Title: Efficacy and Safety of DEH113 in the Treatment of Menstrual Cramp Pain Associated With Primary Dysmenorrhea
Acronym: LIBERTÀ
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEH113-III-0123
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEH113 (Experimental): The patient must take two (2) DEH113 tablets, if pain, up to three times a day.
  Interventions: Drug: DEH113
- Control (Placebo Comparator): The patient must take two (2) DEH113 placebo tablets, if pain, up to three times a day.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: DEH113 — Tablets
  Arms: DEH113
Drug: Placebo Comparator — Tablets
  Other Names: Placebo
  Arms: Control

SUMMARY:
The purpose of this study if to evaluate the efficacy and safety of DEH113 in the Treatment of Menstrual Cramp Pain Associated With Primary Dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent to participate in the study prior to admission to the study;
* Female patients aged between 16 and 35 years old, inclusive;
* History of regular menstrual cycles, occuring between every 21 to 35 days;
* Clinical history compatible with the diagnosis of primary dysmenorrhea;
* Self-reported history of ≥ 4 painful cycles, with moderate or severe menstrual cramps, in the six (06) months prior to selection for the study.

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea;
* History of non-response to treatment with non-steroidal anti-inflammatory drugs (NSAIDs) to relieve menstrual cramps;
* Onset of primary dysmenorrhea after starting to use oral contraceptives;
* Use of oral contraceptives for < 4 months prior to study selection;
* Use of an intrauterine device (IUD), hormonal implants or contraceptive injections in the last six (06) months;
* Previous diagnosis or physical examination findings and/or clinical and/or surgical history that may indicate the presence of endometriosis, pelvic inflammatory disease, adenomyosis, mullerian duct malformation, uterine fibroma, cystic ovary and/or pelvic varicocele;
* History of recurrent pelvic and/or lower abdominal pain outside the menstrual period;
* Presence of known allergy or hypersensitivity to the components of the drugs used during the clinical trial;
* History of hypersensitivity reactions, such as asthma attacks or other types of allergic reactions, to acetylsalicylic acid or other NSAIDs;
* Previous diagnosis of glaucoma;
* Previous diagnosis of kidney and/or liver failure;
* Presence of blood dyscrasias and situations of bone marrow suppression;
* Diagnosis of acute intermittent hepatic porphyria;
* Diagnosis of congenital deficiency of glucose-6-phosphate dehydrogenase (G6PD);
* Presence of mechanical stenosis in the gastrointestinal tract;
* Previous diagnosis of paralytic ileus or intestinal atony
* Diagnosis of myasthenia gravis;
* Previous diagnosis of severe ulcerative colitis or toxic megacolon complicated with ulcerative colitis
* Participants with a history of alcohol or illicit drug use disorder in the last two (02) years;
* Participants with a current medical history of cancer and/or cancer treatment in the last five (05) years;
* Any finding of clinical observation (clinical/physical evaluation) or laboratory condition that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical trial or presence of uncontrolled chronic disease(s);
* Participants who are pregnant, nursing or planning to become pregnant;
* Disagreement with the use of a known effective barrier contraceptive method, unless using a stable oral contraceptive for three months or more (which must be maintained throughout the study), or surgically sterile or who expressly declare themselves exempt from risk of pregnancy for not exercising sexual practices or exercising them in a non-reproductive manner;
* Participation in a clinical research protocol in the last 12 months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator judges that there may be a direct benefit to it;

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women with moderate to severe pain associated with primary dysmenorrhea.
Enrollment: 78 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Sum of Total Pain Relief (TOTPAR) over 0-6 hours post-dose | 6 hours post-dose
  Pain relief will be evaluated considering the Sum of Total Pain Relief (TOTPAR) over 0-6 hours post-dose. Pain relief will be evaluate using a Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief).

SECONDARY OUTCOMES:
Sum of Total Pain Relief (TOTPAR) over 0-4 and 0-8 hours post-dose | 4 and 8 hours post-dose
  Pain relief will be evaluated considering the Sum of Total Pain Relief (TOTPAR) over 0-4 and 0-8 hours post-dose. Pain relief will be evaluate using a Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief).
Sum of Pain Intensity Difference (SPID) over 4, 6 and 8 hours post-dose. | 4, 6 and 8 hours post-dose
  Sum of Pain Intensity Difference (SPID) over 4, 6 and 8 hours post-dose. The pain intensity will be assessed using a Categorical 4-point scale (0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain).
Use of rescue medication | 24 hours post-dose
  Proportion of participants who used rescue medication in the first 24 hours after the first drug intake, amount of rescue medication used in the first 24 hours after the first drug intake, and time elapsed between the last drug intake and the first administration of rescue medication.
Number of additional drug intake | 24 hours post-dose
  Number of additional drug intake during the 24 hours after the first drug intake
Patients' Global Impression of Change (PGIC) | 8 hours post-dose
  Patients' Global Impression of Change (PGIC) will be assessed after 8 hours post-dose or immediately before the intake of rescue medication.
Incidence of Adverse Events Associated with DEH113 in the Treatment of Primary Dysmenorrhea | 7 days post dose
  The safety will be evaluated considering the incidence of adverse events (AEs) reported during the study period.

IPD SHARING:
Plan to Share IPD: No